CLINICAL TRIAL: NCT00162916
Title: A Randomized Controlled Trial of Antidepressant Maintenance for Major Depression Following Mild Traumatic Brain Injury
Brief Title: Antidepressant Maintenance in Traumatic Brain Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ontario Neurotrauma Foundation (Other)
Responsible Party: Mark J Rapoport, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rapoportm-ONF2004-abi-dep-03
Record Dates: First submitted 2005-09-10; First posted 2005-09-13 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Depression
Keywords: Traumatic Brain Injury; Depression; Antidepressant medication; Double-Blind Study; Brain Injuries; Antidepressive Agents; Citalopram; Double-Blind Method
MeSH Terms: conditions — Depression; Brain Injuries, Traumatic; Brain Injuries | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: citalopram

INTERVENTIONS:
Drug: citalopram — 20mg or 40mg, once daily, for 40 weeks
  Other Names: Celexa
  Arms: 2
Drug: Placebo — Cornstarch
  Arms: 1

SUMMARY:
The purpose of the study is to explore to what extent continuing the antidepressant medication citalopram (Celexa), after depression has responded to treatment, helps prevent the return of depressive symptoms in patients with recent traumatic brain injury (TBI).

DETAILED DESCRIPTION:
While antidepressants are effective in treating major depression following TBI, there is a lack of certainty as to how long antidepressants must be continued following improvement of symptoms. Many studies published in the last decade strongly show that antidepressants prevent relapse in patients with major depression in the absence of traumatic brain injury (TBI). However, is it unknown as to whether this is the case following TBI. The aim of this study is to determine whether being on an antidepressant for a year reduces the risk of relapse of depression.

Patients diagnosed with major depression following mild TBI will be treated for ten weeks with the antidepressant drug citalopram. Those who respond, meaning that the symptoms of depression have lessened significantly, will be randomly assigned to either continue taking the citalopram for one year or to take a placebo for one year. Every four weeks, for an additional forty weeks, patients will be assessed for relapse of depression. This study will have a double-blind design, meaning that neither patient nor clinician know whether citalopram or placebo is being administered.

The primary outcome of interest will be a comparison of the percentage of patients who have a recurrence of major depression while continued on citalopram compared with those who were switched to placebo after the acute phase. Recurrence will be defined as meeting Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for major depression and a Hamilton Depression Scale (HAM-D) score of > 16. Or meeting DSM-IV criteria for major depression and having a Clinical Global Impression (CGI) severity score of >= 4 and a CGI illness score of >= 3. The HAM-D and CGI will be administered every four weeks for forty weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* TBI within the last year (this is consistent with clinic population)
* Mild TBI
* Written, informed consent
* Diagnosis of major depressive episode using the depression module of the Structured Clinical Interview for DSM-IV Axis I disorders (SCID-IV), and baseline 17-item Hamilton Depression (HAM-D) Rating Scale score of 16 and above (prior to selective serotonin reuptake inhibitor [SSRI] treatment)
* Response to citalopram 20 or 40mg/d, as defined as a reduction in baseline HAM-D of >= 50%, and HAM-D score of 10 or below; or response to citalopram defined as not meeting DSM-IV criteria for major depression and Clinical Global Impression - severity of mildly ill, borderline ill, or normal and a Clinical Global Impression - improvement of much improved or very much improved impression.

Exclusion Criteria:

* Prior TBI or other focal brain disease (e.g., stroke, tumour)
* Significant acute medical illness including: drug overdose; severely disturbed liver, kidney, lung or heart function; anemia; hypothyroidism; uncontrolled diabetes; Parkinson's disease; Huntington's chorea; progressive supranuclear palsy; brain tumor; subdural hematoma; or multiple sclerosis.
* Current alcohol or substance abuse
* A brain computed tomographic (CT) scan revealing focal lesions that could not be interpreted as consistent with TBI
* Presence of premorbid psychiatric diagnosis of schizophrenia, dementia or bipolar disorder
* Prior episode of major depression in two years prior to TBI, based on SCID-IV interview
* Prior treatment with citalopram or contraindications to receiving treatment with citalopram

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-05; Primary Completion 2008-05 (Actual); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
recurrence of major depression by administering the Hamilton Depression Rating Scale (HAM-D) and Clinical Global Impressions Scale (CGI) every 4 weeks for 40 weeks | 40 weeks

SECONDARY OUTCOMES:
general cognitive function at baseline, 10 weeks and on termination of the trial | 40 weeks
list of adverse drug events at baseline, 10 weeks and on termination of the trial | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Rapoport, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Rapoport MJ, Mitchell RA, McCullagh S, Herrmann N, Chan F, Kiss A, Feinstein A, Lanctot KL. A randomized controlled trial of antidepressant continuation for major depression following traumatic brain injury. J Clin Psychiatry. 2010 Sep;71(9):1125-30. doi: 10.4088/JCP.09m05086blu. Epub 2010 Apr 20. PMID 20441723
- See also: Ontario Neurotrauma Foundation - funding agency for this study — http://www.onf.org